CLINICAL TRIAL: NCT03804814
Title: Assessing a Model for Hepatitis C Elimination: Measuring Patient and Health System Outcomes After Motivational Interviewing Interventions to Increase Treatment Engagement
Brief Title: Motivational Interviewing for HCV Elimination
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pandemic impacted ability to recruit and enroll
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Lisa Barrett, Assistant Professor, Dalhousie University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SAIL-003
Record Dates: First submitted 2018-12-06; First posted 2019-01-15 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Hepatitis C
Keywords: Motivational Interviewing; Healthcare delivery
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing Training (Active Comparator): Health care providers will be trained in motivational interviewing for use in Hepatitis C patient encounters.
  Interventions: Behavioral: Motivational Interviewing Training
- Standard Clinical Encounter (No Intervention): Health care providers will not be trained in motivational interviewing for use in Hepatitis C patient encounters.

INTERVENTIONS:
Behavioral: Motivational Interviewing Training — Motivational Interviewing is a directive, client-centered counselling style intended to elicit behavior change by helping patients reach health goals through their own desires and actions.
  A certified and experienced Motivational Interviewing trainer will develop and deliver the curriculum to healthcare providers.
  Arms: Motivational Interviewing Training

SUMMARY:
This study addresses a difficult barrier to hepatitis C elimination, specifically development and maintenance of a productive relationship between the health care provider and patient to ensure both treatment success and engagement in harm reduction services. Improvements in these domains may be observed through the use of a technique called "Motivational Interviewing" (MI). The aim of this study is to determine whether a customized motivational interviewing curriculum by general primary care and addictions medicine primary care providers changes rates of curative hepatitis C therapy completion.

ELIGIBILITY:
Patient Inclusion Criteria:

* Willingness to participate and provide informed consent
* Positive HCV RNA Result
* ≥18 years of age

Patient Exclusion Criteria:

* Unwilling or unable to provide consent

Health Care Provider Inclusion Criteria:

* Willingness to participate and provide informed consent
* Has a hepatitis C care experience

Health Care Provider Exclusion Criteria:

* Unwilling or unable to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
HCV Treatment Completion | Through study completion, an average of 2 years
  To measure the number of patients who complete HCV therapy

SECONDARY OUTCOMES:
Time from care engagement to treatment initiation | Through study completion, an average of 2 years
Number of unique Hepatitis C related and unrelated health system visits | Through study completion, an average of 2 years
Number of scheduled and attended medical care appointments | Through study completion, an average of 2 years
Self-reported intent to initiate and maintain HCV treatment assessed by questionnaire | Through study completion, an average of 2 years
Healthcare provider knowledge, attitudes, and behavior about motivational interviewing and training assessed by questionnaire | Through study completion, an average of 2 years
Time to complete prescribed HCV treatment course | Through study completion, an average of 2 years
Percentage of eligible individuals that initiate HCV therapy | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No